CLINICAL TRIAL: NCT05170776
Title: Efficacy of Adding Pilates to Postural Correction Exercise on Nerve Root Function and Electromyography Activity in Symptomatic Forward Head Posture: Randomized Controlled Trial
Acronym: FHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003411
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Forward Head Posture
Keywords: forward head psture; Pilates exercise; postural correction exercise; nerve root function
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: this trial has three groups; one experimental and two groups control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates and postural correction exercise (Experimental): pilates and postural correction exercise will be received three times a week for 10 weeks
  Interventions: Other: Pilates and postural correction exercise
- Pilates exercises (Active Comparator): pilates exercise will be received three times a week for 10 weeks
  Interventions: Other: Pilates exercises
- postural correction exercises (Active Comparator): postural corrections exercise will be received three times a week for 10 weeks
  Interventions: Other: postural correction exercises

INTERVENTIONS:
Other: Pilates and postural correction exercise — ten exercises will be performed:
  1. Hip Twist Level 1
  2. Double leg stretch Level 1
  3. Double leg stretch Level 2
  4. One leg stretch Level 1
  5. Clam Level 1
  6. Scissors Level 1
  7. Arm openings Level 1
  8. Breast stroke prep Level 1t
  9. Hip Twist Level 1.
  10. Breast stroke prep Level 2 as for level 1 postural correction exercise
  1-Strengthening deep cervical flexors 2-Stretching cervical extensors 3- Strengthen shoulder retractors 4-Unilateral and bilateral pectoralis stretch
  Arms: Pilates and postural correction exercise
Other: Pilates exercises — ten exercises will be performed:
  1. Hip Twist Level 1
  2. Double leg stretch Level 1
  3. Double leg stretch Level 2
  4. One leg stretch Level 1
  5. Clam Level 1
  6. Scissors Level 1
  7. Arm openings Level 1
  8. Breast stroke prep Level 1t
  9. Hip Twist Level 1.
  10. Breast stroke prep Level 2 as for level 1
  Arms: Pilates exercises
Other: postural correction exercises — postural correction exercise in the form of :
  1. Strengthening deep cervical flexors through chin tucks,
  2. Stretching cervical extensors through a chin drop
  3. Strengthen shoulder retractors
  4. Unilateral and bilateral pectoralis stretch alternating each two-week period.
  Arms: postural correction exercises

SUMMARY:
to investigate the Efficacy of adding Pilates to postural correction exercise on nerve root function and electromyography activity in symptomatic forward head posture: Randomized Controlled Trial

DETAILED DESCRIPTION:
Forward head posture (FHP) is nowadays the most common postural problem. In FHP, the head protrudes forward from the sagittal plane and appears to be positioned in front of the body, and this condition is considered the most common postural deformity. The prevalence of anterior head translation in neck pain patients was found to be 37%, out of which 58% were females and 42%were males. FHP is among the most common abnormal postures in upper quarter. 85% of patients with myofascial pain syndrome have FHP. Even more alarming is how frequently these problems are seen in younger populations since it's suggested that problems at a young age may lead to more serious consequences later in life. Pilate's method is a physical fitness system that was developed during the First World War in the early 20th century by Joseph Hubertus Pilates. Direction Control and Range Control exercises are two key types of specific exercises that should be used when specific uncontrolled movements are found. Pilates is a mind-body exercise that focuses on strength, core stability, flexibility, muscle control, posture and breathing. Exercises can be mat-based or involve use of specialized equipment. Six major components of Pilates as: Centering, Concentration, Control, Precision, Flow and Breathing.

pilates exercise and postural correction play a major role in restoring the normal posture in patients with forward head posture so this trial will be conducted to investigate efficacy of adding Pilates to postural correction exercise on nerve root function and electromyography activity in symptomatic forward head posture.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 20-45 years old with symptomatic forward head posture will be included in this study
* Participants have FHP if CVA ≤ 50 Non- athletes
* Normal body mass index (BMI) (18- 24.9). (BMI = body mass in kg divided by subject height in meters).

Exclusion Criteria:

* any spinal problems
* Temporomandibular disease
* Participants with experience in pilates and who will not be sedentary were excluded from the study
* Previous surgery in the neck and shoulder
* neurological symptoms of the upper extremities during screening tests (e.g., Spurling test and upper limb tension tests)
* red flags suggesting of cancer, infection, vascular insufficiency
* Cervical radiculopathy or mylopathy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
nerve root function | up to ten weeks
  nerve root function in the form of somatosensory evoked potential will be measure by electromyograph.

SECONDARY OUTCOMES:
pain intensity | up to ten weeks
  pain intensity will be measure by visual analogue scale.
neck disability | up to ten weeks
  neck disability will be measure by Arabic neck disability index
flexion and extension endurance test | up to ten weeks
  the endurance will be measured by stop watch
muscle amplitude | up to ten weeks
  electromyography will be used to measure the muscle amplitude in the form of root mean square
craniovertebral angle | up to ten weeks
  craniovertebrel angle will be measured by surgimap program

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt